CLINICAL TRIAL: NCT03872414
Title: Emotion Study (Improving Neural Dysregulation in Advanced Age: A Neurofeedback Approach)/Substudy: Flexible Brain Study
Brief Title: Emotion Study/Substudy: Flexible Brain Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Florida Department of Health (Other Government); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: IRB201300814-PD -N; 1R21AG057200 (NIH); UL1TR001427 (NIH); 20A15 (Other: Ed and Ethel Moore Alzheimer's Disease Research Program)
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Aging; Emotions; Parkinson Disease
Keywords: Emotional Aging; Neurofeedback
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy Younger Group (Experimental): Participants will receive rt-fMRI training to increase anterior cingulate cortex activation.
  Interventions: Behavioral: Anterior cingulate cortex activation
- Healthy Older Group (Experimental): Participants will receive rt-fMRI training to increase anterior cingulate cortex activation.
  Interventions: Behavioral: Anterior cingulate cortex activation
- Parkinson Disease Group (Experimental): Participants will receive rt-fMRI training to increase anterior cingulate cortex activation.
  Interventions: Behavioral: Anterior cingulate cortex activation
- Control Group (Active Comparator): Participants will receive rt-fMRI training to increase primary auditory cortex activation.
  Interventions: Behavioral: Primary auditory cortex activation

INTERVENTIONS:
Behavioral: Anterior cingulate cortex activation — Functional Magnetic Resonance Imaging Participants in the experimental group will be trained using functional magnetic resonance imaging to regulation brain activity in anterior cingulate cortex.
  The anterior cingulate cortex is a brain region that is known to be involved in emotion processing. Activation of this region is expected to improve emotion processing.
  Arms: Healthy Older Group; Healthy Younger Group; Parkinson Disease Group
Behavioral: Primary auditory cortex activation — Functional Magnetic Resonance Imaging Participants in each group will be trained using functional magnetic resonance imaging to regulation brain activity in primary auditory cortex. The primary auditory cortex is a brain region that is NOT specifically involved in emotion processing. Activation of this region is NOT expected to improve emotion processing; and thus activation of this brain region serves as "control/placebo" condition in the current design (placebo comparator).
  Arms: Control Group

SUMMARY:
The proposed research applies the highly innovative technology of real-time functional Magnetic Resonance Imaging (rtfMRI) to examine plasticity of brain-regulatory mechanisms related to cognitive and affective processing and to determine benefits for cognition and affect in young and older adults and in Parkinson Disease (PD) patients.

DETAILED DESCRIPTION:
There is increasing evidence that age-related alterations in brain function associated with affective processing and attention contribute to these motivational and emotional changes with age.

Based on these theoretical considerations as well as the previous study's data, the proposed research will apply well-tested emotion processing and attention paradigms to address the pivotal question of whether brain activity can be modulated in healthy aging and PD (in the substudy) via contingent rt-fMRI neurofeedback and whether this neuroregulatory modulation increases emotion processing and cognitive performance.

ELIGIBILITY:
Inclusion Criteria: Young adults

* aged 18-35 years of age
* native English speaker
* at least 8th grade education
* generally physically and neurologically healthy as determined by the Health Demographics Screener
* eligible for MRI as determined by the MRI Eligibility Interview (including not being pregnant)
* scores within normal limits on a cognitive screener (MoCA)
* no indication of serious psychiatric disturbance including major depression (based on Mental Health Screener)
* willing and able to give informed consent

Inclusion Criteria: Older adults

* age 55-100 years of age
* native English speaker
* at least 8th grade education
* generally physically and neurologically healthy as determined by the Health Demographics Screener
* eligible for MRI as determined by the MRI Eligibility Interview
* no indication of dementia based on score of 30 or above on the Telephone Interview for Cognitive Status and nonimpaired score on the Montreal Cognitive Assessment (MoCA -- score of 22 and above)
* no indication of serious psychiatric disturbance including current major depression (based on Mental Health Screener)
* willing and able to give informed consent

Inclusion Criteria: Parkinson patients

* must meet criteria for diagnosis of idiopathic Parkinson disease according the UK Brain Bank by a movement trained neurologist.
* age 55-100 years of age
* native English speaker
* at least 8th grade education
* generally physically and neurologically healthy other than Parkinson disease
* eligible for MRI as determined by the MRI Eligibility Interview
* no indication of dementia based on cognitive screening measures (TICS -- score of 30 or above, and MoCa -- score of 22 and above)
* no indication of serious psychiatric disturbance including current major depression
* willing and able to give informed consent

Inclusion Criteria: Individuals with SCD and a family history of dementia or Alzheimer's disease

* age 55-100 years of age
* native English speaker
* at least 8th grade education
* generally physically and neurologically healthy as determined by the Health Demographics Screener
* eligible for MRI as determined by the MRI Eligibility Interview
* no indication of dementia based on score of 30 or above on the Telephone Interview for Cognitive Status and nonimpaired score on the Montreal Cognitive Assessment (MoCA -- score of 22 and above)
* no indication of serious psychiatric disturbance including current major depression (based on Mental Health Screener)
* willing and able to give informed consent
* community-dwelling with subjective report of cognitive complaints with scores >16 on the Cognitive Change Index (CCI-20)
* no evidence of dementia or mild cognitive impairment based on cognitive screening using the MoCA; scores must fall within normal limits for age, education, and sex
* no psychometric evidence of neuropsychological impairment on a modified Neuropsychological Battery from the NACC Unified Data Set, version 3
* score of 0 on the Global Clinic Dementia Rating (CDR) scale
* normal functional behavior in terms of daily activities, based on the Functional Activities Scale (FAQ)
* availability of an informant (over the phone) who can provide information about the participant's complaints using the informant version of the CCI-20, and corroborate normal activities of daily living on the FAQ and the CDR scale.

Exclusion Criteria:

* Pregnant or possibly pregnant
* Claustrophobia
* Large pieces of metal in the body, particularly in the face and neck.
* Piercings or metal implants that cannot be removed from the body
* Surgery on the brain or any prior serious brain damage or disease
* Dementia or severe cognitive disorders
* use of antipsychotics, sedatives, or other medications with significant anticholinergic properties (due to potential influence on memory)
* use of prescribed 'memory enhancing' medications such as Aricept or Namenda.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Change in BOLD signal response | Baseline; Day 8
  Change in blood-oxygen-level dependent (BOLD) signal response of the anterior cingulate cortex.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Ebner, PhD, Principal Investigator — University of Florida, Department of Psychology
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No